CLINICAL TRIAL: NCT02196558
Title: A Phase 1/2 Study of Repeated Subcutaneous E6011 Administration in Japanese Subjects With Rheumatoid Arthritis
Brief Title: A Study of E6011 in Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E6011-J081-103
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2017-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Japanese subjects
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — quetmolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- E6011, 100 mg Arm (Experimental): E6011 will be administered repeatedly, subcutaneously at Week 0, 1, 2, followed by every 2 weeks upto 10 weeks (treatment phase).100 mg group will receive E6011 subcutaneously, 1 ml. If a subject intends to continue administrations; the subject will receive a total of 20 subsequent biweekly administrations (40 weeks) at stable dose (Extension phase).
  Interventions: Drug: E6011
- E6011, 200 mg Arm (Experimental): E6011 will be administered repeatedly, subcutaneously at Week 0, 1, 2, followed by every 2 weeks upto 10 weeks (treatment phase). 200 mg group will receive E6011 subcutaneously, 1 ml each at two sites. If a subject intends to continue administrations; the subject will receive a total of 20 subsequent biweekly administrations (40 weeks) at stable dose (Extension phase).
  Interventions: Drug: E6011
- E6011, 400 mg Arm (Experimental): E6011 will be administered repeatedly, subcutaneously at Week 0, 1, 2, followed by every 2 weeks up to 10 weeks (treatment phase). 400 mg group will receive E6011 subcutaneously, 1 ml each at four sites or 2 ml each at two sites. If a subject intends to continue administrations, the subject will receive a total of 20 subsequent biweekly administrations (40 weeks) at stable dose (Extension Phase).
  Interventions: Drug: E6011

INTERVENTIONS:
Drug: E6011

SUMMARY:
This study consist of treatment phase (12 weeks) and extension phase (40 weeks). This study is a multicenter, open-label, uncontrolled, multiple ascending dose (MAD) study to evaluate mainly the safety and tolerability of 12-week repeated subcutaneous administration of E6011 in Japanese subjects with Rheumatoid Arthritis. First 12 subjects will enroll as 100 mg group, next 12 subjects will enroll as 200 mg group, and last 9 subjects will enroll as 400 mg group. A total of 33 subjects will receive repeated subcutaneous administration of E6011. Subjects who roll over onto the Extension phase will have continued monitoring until 52 weeks after the initial administration.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Japanese patients aged 20 to 64 years old at the time of informed consent.
2. Diagnosed with rheumatoid arthritis (RA) who meet the 1987 ACR or 2010 ACR/EULAR criteria.
3. Presenting tenderness in more than 4 joints (out of 68) and swelling in more than 4 joints (out of 66) at Screening and Observation phase.
4. Never been treated with non-anti-TNF biologics or never been treated with 2 or more anti-TNF agents.
5. Subjects with greater than or equal to 0.6 mg/dL of high-sensitivity CRP (hs-CRP) level or greater than or equal to 28 mm/hr of erythrocyte sedimentation rate (ESR) at Screening.
6. Weighs greater than or equal to 30 kg and less than or equal to 100 kg at Screening.
7. Consent to use contraception (both the subject and the subject's partner), for at least 70 days after the last dose of study medication starting on the day of informed consent, if the subject is a man capable of reproduction or a woman of childbearing potential.
8. Has voluntarily consented, in writing, to participate in this study
9. Has been thoroughly briefed on the conditions for participation in the study, and is willing and able to comply with all aspects of the protocol.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Any history or complication of inflammatory arthritic disorder other than rheumatoid arthritis or Sjogren's syndrome.
2. Meet Class 4 with the Steinbrocker functional classification.
3. History or current clinical condition, or associated complications of malignant tumor, lymphoma, leukemia, or lymphoproliferative disease.
4. Immunodeficiency or history of HIV infection
5. Infection requiring hospitalization or intravenous administration of antibiotics within 4 weeks before the first dose of study treatment, or an infection requiring oral antibiotics within 2 weeks before the first dose of study treatment.
6. History of tuberculosis or current complication of active tuberculosis.
7. History of severe allergy (shock, or anaphylactoid symptoms).
8. History of clinically important vascular edema, hematemesis, hemorrhagic stool, or hemoptysis.
9. History of acute myocardial infarction, cerebral infarction, cerebral hemorrhage, or arteriosclerosis obliterans.
10. History of clinically important vasculitis (such as mononeuritis multiplex).
11. Tested positive for any of the following at Screening: human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B virus core antibody (HBc antibody), hepatitis B virus DNA (HBV DNA), hepatitis C virus antibody (HCV antibody), human T-lymphotrophic virus Type I antibody (HTLV-1 antibody), or syphilis.
12. Any result other than negative in tuberculosis test (T-SPOT.TB Test or QuantiFERON TB Gold Test) at Screening.
13. Findings indicating a history of tuberculosis on chest X-ray at Screening.
14. Ineligible to participate in the study in the opinion of the investigator or sub investigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (12):
  - Kitakyushu, Fukuoka
  - Sapporo, Hokkaido
  - Kakogawa, Hyōgo
  - Katō, Hyōgo
  - Kahoku-gun, Ishikawa-ken
  - Yokohama, Kanagawa
  - Hamamatsu, Shizuoka
  - Chuo-Ku, Tokyo
  - Meguro-Ku, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-Ku, Tokyo
  - Miyazaki

REFERENCES:
- [Derived] Tanaka Y, Takeuchi T, Umehara H, Nanki T, Yasuda N, Tago F, Kawakubo M, Kitahara Y, Hojo S, Kawano T, Imai T. Safety, pharmacokinetics, and efficacy of E6011, an antifractalkine monoclonal antibody, in a first-in-patient phase 1/2 study on rheumatoid arthritis. Mod Rheumatol. 2018 Jan;28(1):58-65. doi: 10.1080/14397595.2017.1337056. Epub 2017 Jul 6. PMID 28681650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in Japan from 26 May 2014 to 13 July 2017. As planned separate pharmacokinetics (PK) parameters are not reported and PK analyses was performed for serum E6011 concentrations. Also as planned, combined data for Treatment Phase and Expansion Phase is reported.
Pre-assignment Details: Total 53 participants were enrolled and screened, of which 16 were screen failures, 37 participants received study drug in 12-week Treatment Phase. Out of them, 32 participants completed 12-week Treatment Phase. Of 32 participants, 28 participants entered Extension Phase, 22 completed 40-week Extension Phase. '>='signifies greater than or equal to.
Groups:
- E6011: 100 mg: Participants received E6011 100 milligram (mg), subcutaneously, injection, at Week 0, 1, 2, followed by every 2 weeks up to Week 10 in Treatment Phase and continued to receive E6011 100 mg, subcutaneously, injection, at every two weeks in Extension Phase (for a total of 52 weeks [Treatment Phase of 12 Weeks and Extension Phase of 40 Weeks]).
- E6011: 200 mg: Participants received E6011 200 mg, subcutaneously, injection, at Week 0, 1, 2, followed by every 2 weeks up to 10 weeks in Treatment Phase and continued to receive E6011 200 mg, subcutaneously, injection, at every two weeks in Extension Phase (for a total of 52 weeks [Treatment Phase of 12 Weeks and Extension Phase of 40 Weeks]).
- E6011: 400 mg: Participants received E6011 400 mg, subcutaneously, injection, at Week 0, 1, 2, followed by every 2 weeks up to 10 weeks in Treatment Phase and continued to receive E6011 400 mg, subcutaneously, injection, at every two weeks in Extension Phase (for a total of 52 weeks [Treatment Phase of 12 Weeks and Extension Phase of 40 Weeks]).
Period: Treatment Phase (12 Weeks)
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg
Started | 12 | 15 | 10
Completed | 12 | 12 | 8
Not Completed | 0 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Participant Choice | 0 | 1 | 1
Not completed — Progression of Disease | 0 | 0 | 1
Period: Extension Phase (40 Weeks)
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg
Started | 11 (Participants who wished to continue, had no safety issues, and had>=20% improvement in joint counts.) | 11 (Participants who wished to continue, had no safety issues, and had>=20% improvement in joint counts.) | 6 (Participants who wished to continue, had no safety issues, and had>=20% improvement in joint counts.)
Completed | 9 | 8 | 5
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Inadequate therapeutic effect | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included group of participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Groups:
- E6011: 100 mg: Participants received E6011 100 mg, subcutaneously, injection, at Week 0, 1, 2, followed by every 2 weeks up to Week 10 in Treatment Phase and continued to receive E6011 100 mg, subcutaneously, injection, at every two weeks in Extension Phase (for a total of 52 weeks [Treatment Phase of 12 Weeks and Extension Phase of 40 Weeks]).
- Total: Total of all reporting groups
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg | Total
Number analyzed (Participants) | 12 | 15 | 10 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (8.95) | 51.5 (12.02) | 48.6 (8.28) | 49.5 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 7 | 29
  Male | 1 | 4 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 15 | 10 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 15 | 10 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to 52 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg
Number analyzed (Participants) | 12 | 15 | 10
Participants
  TEAEs | 10 | 14 | 7
  SAEs | 1 | 3 | 1

2. Secondary Outcome: Number of Participants With Positive Anti-E6011 Antibodies Results
Time Frame: Up to 52 weeks
Population: The safety analysis set included group of participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. Here, "number analyzed" signifies the participants who were evaluable for this outcome measure for given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg
Number analyzed (Participants) | 12 | 15 | 10
Participants
  Treatment Phase (12 Weeks) | 9 | 6 | 1
  Extension Phase (40 Weeks): number analyzed (Participants) | 11 | 11 | 6
  Extension Phase (40 Weeks) | 9 | 5 | 2

3. Secondary Outcome: Serum Concentrations of E6011
Time Frame: At Week 0 (predose), Week 1, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 (postdose)
Population: The pharmacokinetics (PK) analysis set included group of participants who received at least 1 dose of study drug and had at least 1 serum E6011 concentration data. Here, "number analyzed" signifies the participants who were evaluable for this outcome measure for given time points.
Measure: Mean (Standard Deviation); unit: mcg/ml (microgram per milliliter)
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg
Number analyzed (Participants) | 12 | 15 | 10
mcg/ml (microgram per milliliter)
  Week 0 (predose) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Week 1: number analyzed (Participants) | 12 | 15 | 9
  Week 1 | 8.12 (3.06) | 20.0 (9.11) | 39.9 (13.6)
  Week 2: number analyzed (Participants) | 12 | 15 | 9
  Week 2 | 15.7 (6.30) | 37.1 (11.9) | 73.9 (20.7)
  Week 4: number analyzed (Participants) | 12 | 14 | 8
  Week 4 | 15.6 (6.75) | 38.8 (16.6) | 80.9 (28.7)
  Week 6: number analyzed (Participants) | 12 | 13 | 8
  Week 6 | 12.5 (6.04) | 34.8 (16.6) | 82.1 (27.9)
  Week 8: number analyzed (Participants) | 11 | 13 | 7
  Week 8 | 12.4 (7.17) | 35.1 (20.4) | 84.1 (31.3)
  Week 10: number analyzed (Participants) | 11 | 12 | 7
  Week 10 | 12.9 (8.20) | 29.2 (11.1) | 90.7 (38.0)
  Week 12: number analyzed (Participants) | 11 | 12 | 7
  Week 12 | 11.6 (7.02) | 31.2 (11.9) | 90.7 (39.7)
  Week 16: number analyzed (Participants) | 9 | 11 | 5
  Week 16 | 14.4 (6.33) | 28.2 (11.2) | 111 (28.1)
  Week 20: number analyzed (Participants) | 9 | 11 | 5
  Week 20 | 14.6 (6.97) | 30.6 (10.9) | 103 (37.6)
  Week 24: number analyzed (Participants) | 9 | 11 | 5
  Week 24 | 13.7 (7.76) | 30.5 (12.6) | 116 (26.0)
  Week 28: number analyzed (Participants) | 9 | 10 | 5
  Week 28 | 13.8 (8.33) | 33.6 (11.6) | 98.3 (31.1)
  Week 32: number analyzed (Participants) | 8 | 9 | 5
  Week 32 | 15.1 (6.25) | 31.4 (12.4) | 106 (30.7)
  Week 36: number analyzed (Participants) | 8 | 9 | 4
  Week 36 | 14.0 (7.23) | 31.6 (13.4) | 108 (32.4)
  Week 40: number analyzed (Participants) | 8 | 8 | 4
  Week 40 | 14.6 (8.90) | 39.2 (11.5) | 113 (30.2)
  Week 44: number analyzed (Participants) | 8 | 7 | 4
  Week 44 | 13.2 (7.56) | 40.4 (15.5) | 112 (37.9)
  Week 48: number analyzed (Participants) | 8 | 7 | 4
  Week 48 | 14.6 (8.43) | 37.5 (19.0) | 111 (32.9)
  Week 52: number analyzed (Participants) | 8 | 7 | 4
  Week 52 | 16.2 (11.2) | 37.0 (12.7) | 111 (41.1)

ADVERSE EVENTS:
Time Frame: Up to 52 Weeks
Description: As planned, combined safety data for E6011 administered in Treatment phase and Extension phase was reported.
Arm/Group | E6011: 100 mg | E6011: 200 mg | E6011: 400 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/12 | 3/15 | 1/10
Other Adverse Events (participants affected / at risk) | 10/12 | 13/15 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E6011: 100 mg (N=12) | E6011: 200 mg (N=15) | E6011: 400 mg (N=10)
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E6011: 100 mg (N=12) | E6011: 200 mg (N=15) | E6011: 400 mg (N=10)
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 5 | 7 | 4
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Gastric infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood beta-D-glucan increased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Candida test positive (Investigations) | 1 | 0 | 0
Cell marker increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No